CLINICAL TRIAL: NCT02505165
Title: A Clinic-Based Interdisciplinary Intervention for Parents of Children With Cancer
Brief Title: Illness Management and Parental Adjustment to Cancer Treatment
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Oklahoma (Other); Oklahoma State University (Other); Dayton Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NR014248
Record Dates: First submitted 2015-06-17; First posted 2015-07-22 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor; Leukemia; Lymphoma; Brain Tumor
Keywords: Intervention; Illness Uncertainty; Childhood Cancer; Solid Tumor; Leukemia; Lymphoma; Brain Tumor; Randomized clinical trial; Parental uncertainty management intervention; Parent; Oncology; Pediatric
MeSH Terms: conditions — Leukemia; Lymphoma; Brain Neoplasms; Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Uncertainty Intervention (Experimental): A pediatric cancer-specific, clinic based, six-module interdisciplinary uncertainty intervention. Modules one through three target uncertainty prevention. Modules four through six target uncertainty responses for situations in which uncertainty cannot be prevented or avoided.
  Interventions: Behavioral: IMPACT
- Education/Support Only (Other): Sessions in this condition aim to provide education on cancer etiology, medical treatments, side effects, potential short- and long-term effects of treatment and resources that are often helpful to parents of children with cancer. Information presented will be based upon, "Young People with Cancer: A Handbook for Parents", a parent resource developed by the National Cancer Institute. Parents will also be provided with relevant educational brochures from COG. Each session will also include a structured set of questions that will facilitate discussion. All ESO interventionists will be trained in non-directive approaches including reflective listening. Content provided in the ESO sessions will offer valuable information to parents without providing the specific skills of the IMPACT.
  Interventions: Other: ESO

INTERVENTIONS:
Behavioral: IMPACT — • The intervention is 6 sessions lasting approximately 45 minutes reviewing ways to help prevent and respond to illness uncertainty. Sessions occur weekly at already scheduled clinic appointments. Interventions will be delivered by a trained interventionist.
  Other Names: Parent Uncertainty Management Intervention
  Arms: Parent Uncertainty Intervention
Other: ESO — This control is 6 sessions lasting approximately 45 minutes providing education on cancer etiology, medical treatments, side effects, potential short- and long-term effects of treatment and resources that are often helpful to parents of children with cancer. Sessions occur weekly at already scheduled clinic appointments. Interventions will be delivered by a trained interventionist.
  Other Names: Education/Support Only
  Arms: Education/Support Only

SUMMARY:
The purpose of this study is to test the efficacy of a clinic-based intervention designed to reduce illness uncertainty for parents of children who have been recently diagnosed with cancer.

DETAILED DESCRIPTION:
The proposed trial will test the efficacy of the parent-focused clinic-based Parent Uncertainty Management Intervention (PUMI) to improve the outcomes of children newly diagnosed with cancer and their parents. Participants will be randomly assigned to receive equivalent doses of either the PUMI or an Education/Support (ESO) group. Theoretically driven by Mishel's model of illness uncertainty, the PUMI will teach parents about uncertainty prevention and management through the use of medically-specific communication, information management, and problem-solving skills via in-clinic sessions and an online portal. Parents and children will complete measures online at baseline, 1-week, and 3-, 6-, and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* The child has been diagnosed with leukemia or lymphoma, malignant solid tumor, or malignant brain tumor
* The child is being treated for cancer and returning to the medical center (CCHMC or OUHSC).
* The child is 18 years of age or younger
* Recruitment occurs within 2-12 weeks post diagnosis
* The parent is responsible for care and is willing to give consent and participate
* The child is willing to give assent or consent and participate (only for children 8 years old and older)
* The parent gives patient permission to participate.
* Parent is fluent in English

Exclusion Criteria:

* The child is experiencing an imminent medical crisis necessitating significant medical intervention
* The child with cancer is determined to be in the terminal phase of illness and/or is receiving end of life care
* The diagnosis is determined to be a relapse or a second malignancy
* The parent is currently being treated for a serious psychiatric disorder, or, evidences mental retardation
* The parent is younger than 18 years of age
* The parent is not English speaking
* The parent is unwilling to give written permission for child participation
* If the patient's treatment visit schedule is too infrequent to meet the study visit timeline requirements

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 279 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Psychosocial Functioning as assessed by the global severity index (GSI) of the symptom checklist 90. | Change in (global severity index) GSI score from baseline to 1-week post-intervention
  indicator of global psychological symptoms
Psychosocial Functioning as assessed by the global severity index of the symptom checklist 90. | Change in GSI score from baseline to 3-month post-intervention
  indicator of global psychological symptoms
Psychosocial Functioning as assessed by the global severity index of the symptom checklist 90. | Change in GSI score from baseline to 6-month post-intervention
  indicator of global psychological symptoms
Psychosocial Functioning as assessed by the global severity index of the symptom checklist 90. | Change in GSI score from baseline to 12-month post-intervention
  indicator of global psychological symptoms

SECONDARY OUTCOMES:
Post-Traumatic Stress Symptoms as assessed by the Impact of Events Scale-Revised (IES-R) | Change in IES-R total score score from baseline to 1-week post-intervention
  Measure of caregiver post-traumatic stress symptoms
Post-Traumatic Stress Symptoms as assessed by the Impact of Events Scale-Revised (IES-R) | Change in IES-R total score score from baseline to 3-month post-intervention
  Measure of caregiver post-traumatic stress symptoms
Post-Traumatic Stress Symptoms as assessed by the Impact of Events Scale-Revised (IES-R) | Change in IES-R total score score from baseline to 6-month post-intervention
  Measure of caregiver post-traumatic stress symptoms
Post-Traumatic Stress Symptoms as assessed by the Impact of Events Scale-Revised (IES-R) | Change in IES-R total score score from baseline to 12-month post-intervention
  Measure of caregiver post-traumatic stress symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ahna LH Pai, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided
Due to the sensitive nature of the measures that provided information on the participants psychologically symptoms the final dataset will be stripped of identifiers prior to any release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics due the relatively rare pediatric oncological diagnoses of the children in the study. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using the highest standards of practice; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Szulczewski L, Mullins LL, Bidwell SL, Eddington AR, Pai ALH. Meta-Analysis: Caregiver and Youth Uncertainty in Pediatric Chronic Illness. J Pediatr Psychol. 2017 May 1;42(4):395-421. doi: 10.1093/jpepsy/jsw097. PMID 28177514
- [Background] Sharkey CM, Schepers SA, Drake S, Pai ALH, Mullins LL, Grootenhuis MA. Psychosocial Risk Profiles Among American and Dutch Families Affected by Pediatric Cancer. J Pediatr Psychol. 2020 May 1;45(4):463-473. doi: 10.1093/jpepsy/jsaa012. PMID 32196095
- [Result] Morrison CF, Szulczewski L, Strahlendorf LF, Lane JB, Mullins LL, Pai AL. Designing Technology to Address Parent Uncertainty in Childhood Cancer. ANS Adv Nurs Sci. 2016 Jan-Mar;39(1):15-25. doi: 10.1097/ANS.0000000000000100. PMID 26836990
- [Result] Marsolo K, Shuman W, Nix J, Morrison CF, Mullins LL, Pai AL. Reducing Parental Uncertainty Around Childhood Cancer: Implementation Decisions and Design Trade-Offs in Developing an Electronic Health Record-Linked Mobile App. JMIR Res Protoc. 2017 Jun 26;6(6):e122. doi: 10.2196/resprot.7523. PMID 28652227
- [Result] Basile NL, Chardon ML, Peugh J, Edwards CS, Szulczewski L, Morrison CF, Nagarajan R, El-Sheikh A, Chaney JM, Pai ALH, Mullins LL. Relationship Between Caregiver Uncertainty, Problem-Solving, and Psychological Adjustment in Pediatric Cancer. J Pediatr Psychol. 2021 Oct 18;46(10):1258-1266. doi: 10.1093/jpepsy/jsab065. PMID 34350968
- [Derived] Nebeker C, Murray K, Holub C, Haughton J, Arredondo EM. Acceptance of Mobile Health in Communities Underrepresented in Biomedical Research: Barriers and Ethical Considerations for Scientists. JMIR Mhealth Uhealth. 2017 Jun 28;5(6):e87. doi: 10.2196/mhealth.6494. PMID 28659258